CLINICAL TRIAL: NCT05940454
Title: Efficacy of Pericapsular Nerve Group Block in the Prevention of Postoperative Pain in Shoulder Surgery
Brief Title: Pericapsular Nerve Group Block in Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, EMİNE ASLANLAR, Assistant professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PENG
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
Keywords: pericapsular nerve group block; postoperative pain; shoulder surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nerve group block (Group P) (Experimental): Pericapsular nerve group block will be performed with 20 ml of 0.5% bupivacaine hydrochloride before general anesthesia is applied to the patients in Group P.
  Interventions: Procedure: Pericapsular nerve group block
- control group (Group C) (No Intervention): No block will be applied to patients in Group C.

INTERVENTIONS:
Procedure: Pericapsular nerve group block — The patient's arm is externally rotated and abducted at 45 degrees. A longitudinal linear ultrasound probe is placed between the coracoid and the humeral head. After defining the humeral head, the tendon of the subscapular muscle and the deltoid muscle on it, a 50 mm needle is inserted with the "in-plane" technique. When the needle passes through the deltoid muscle and touches the subscapularis tendon, a hard bone-like tissue is felt and the needle is not advanced any further. It is noteworthy that the subscapularis tendon is very rigid and resistant to needle penetration when performing the pericapsular nerve group block. The needle tip is placed between the deltoid muscle and the subscapularis tendon and a local anesthetic drug (20 ml, %0.5 bupivacain hydrochlorur) is injected
  Arms: Pericapsular nerve group block (Group P)

SUMMARY:
Dear Patient, You have been scheduled for shoulder surgery by your surgeon. This surgery is performed under general anesthesia, that is, by putting the patient to sleep, and then moderate or severe pain is experienced. In order to prevent this post-operative pain, painkillers are given through the vascular access or the operated area, namely the shoulder, is locally anesthetized. Many techniques are used to numb the shoulder locally. One of these techniques is the pericapsular nerve group block and it is a newly defined technique.

In this block, some of the nerves that carry the pain sensation of the shoulder are temporarily anesthetized with local anesthetics.

This study will investigate how effective this block is in reducing pain associated with shoulder surgery.

DETAILED DESCRIPTION:
Dear Patient, You have been scheduled for shoulder surgery by your surgeon. This surgery is performed under general anesthesia, that is, by putting the patient to sleep, and then moderate or severe pain is experienced. In order to prevent this pain to be experienced, analgesics are given through the vascular access or the operated area, namely the shoulder, is locally anesthetized. Different techniques are used to numb the shoulder locally. One of these techniques is pericapsular nerve group block. In this block, some of the nerves that carry the pain sensation of the shoulder are temporarily anesthetized with local anesthetics. Thus, it is aimed to reduce post-operative pain.

In this study, we plan to investigate how effective the pericapsular nerve group block is on postoperative pain. In this scientific study, patients will be randomly divided into two groups. Pericapsular nerve group block will be applied to one group of patients, while the other group will not be blocked. Pain medication will be administered intravenously to both groups before waking them up, and at the same time, a device called 'Patient Controlled Analgesia' (PCA) containing a very strong pain medication will be inserted in all patients in the service.

This device; It is a device that contains analgesics and gives analgesics to the patient through the vascular access according to the patient's request, and it works with the help of a button on it. When the patient feels pain, he will press the button and the device will give the medicine to the patient in a predetermined dose and time. The device records the total amount of pain medication sent in 24 hours on its screen. The amount of medication delivered by this device will be compared between patients with and without block. Thus, the effect of pericapsular nerve group block on postoperative pain will be investigated.

What are the procedures to be applied in the research? The surgery that will be applied to you is performed under general anesthesia. Pericapsular nerve group block, which is one of the pain relief methods we apply for shoulder surgery; It involves administering a local anesthetic drug with the help of a needle between the muscles in the shoulder and numbing your shoulder area.

After the blocking procedure, painful stimulus will be given and it will be checked whether you have pain and loss of sensation and what it is worth. If there is loss of feeling, the block will be considered successful.

After the evaluation of the block procedure is completed, you will be given general anesthesia, that is, you will be put to sleep. At the end of the surgery and at the 4th, 8th, 12th and 24th hours after the surgery, the severity of your pain will be evaluated and the total amount of analgesic consumed will be recorded. A scale that includes scoring pain between 0 and 10, called "NRS (numerical rating scale)" will be used. With this scale, you will be asked to give a score between 0 and 10 according to the severity of the pain. 0 points; "no pain", 5 points; moderate pain, and 10 points means "the most severe pain the patient has ever felt".

ELIGIBILITY:
Inclusion Criteria:Patients scheduled for elective arthroscopic shoulder surgery under general anesthesia Patients aged 18 to 65 years American Society of Anesthesiologists (ASA) physical status value I-III patients

-

Exclusion Criteria:

* coagulopathy,
* neuropathy,
* use of anticoagulants,
* severe diabetes mellitus,
* local anesthetic and/or opioid allergy or sensitivity,
* a history of chronic pain,
* pre-existing psychiatric illness,
* can't understand pain scoring,
* Body mass index greater than 35 kg/m2,
* There is an infection in the body area to be blocked,
* Continuing follow-up and treatment in the intensive care unit,
* open shoulder surgery
* do not approve the informed consent form
* pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the effect of pericapsular nerve group block on postoperative pain. | 24 hours
  Postoperative pain will be assessed using the NRS score (Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain) at 0, 4, 8, 12, and 24 hours.

SECONDARY OUTCOMES:
Postoperative pain assessment is to evaluate time to first analgesia requirement, total amount of analgesic consumed, and complications. | 24 hours
  Demanded/administered analgesic ratio in PCA (patient control analgesia) device

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263
- [Background] Ramadurai R, Bhoi D, Nagarajappa A, Amar P. Pericapsular nerve group block (PENG) at neutral position for shoulder manipulation: A feasible approach for a new indication. J Clin Anesth. 2021 Dec;75:110541. doi: 10.1016/j.jclinane.2021.110541. Epub 2021 Oct 12. No abstract available. PMID 34653775